CLINICAL TRIAL: NCT04519424
Title: A Phase 2, Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate CSL324 in Coronavirus Disease 2019 (COVID-19)
Brief Title: CSL324 in COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business reasons, not safety issues.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL324_COVID-19
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSL324 (Experimental): CSL324 administered intravenously
  Interventions: Biological: CSL324
- Placebo (Placebo Comparator): Normal saline administered intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL324 — Recombinant anti-granulocyte colony-stimulating factor (G-CSF) receptor monoclonal antibody
  Arms: CSL324
Drug: Placebo — Normal saline (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
This is a phase 2, prospective, multicenter, randomized, double blind, placebo controlled, parallel group study to evaluate the safety and efficacy of intravenous (IV) administration of CSL324, administered in combination with SOC treatment, in subjects with COVID 19.

For the purposes of this study, standard of care (SOC) may include any written or established treatment protocol followed at the study site for the treatment of severe COVID-19 or its complications, including off-label use of marketed pharmaceutical products and / or products with emergency use authorization granted for the treatment of COVID-19 (ie, not yet marketed) (eg, remdesivir).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time informed consent is obtained
* Positive for SARS-CoV-2 infection determined by a diagnostic test approved by the Food and Drug Administration (FDA) or allowed under an emergency use authorization
* Chest computed tomography (CT) scan or X ray results confirming interstitial pneumonia
* Meets ≥ 1 of the following criteria (subjects improving while on respiratory support still qualify):

  * Respiratory rate > 30 breaths per minute
  * Peripheral (capillary) oxygen saturation (SpO2) ≤ 93% on room air
  * Partial pressure of oxygen in arterial blood (PaO2) to fraction of inspired oxygen (FiO2) ratio (PaO2 / FiO2) < 300
  * SpO2 / FiO2 ratio < 218 (if PaO2 / FiO2 ratio is not available)
  * Radiographic lung infiltrates > 50%

Exclusion Criteria:

* Currently enrolled, planning to enroll, or participated, within the last 30 days, in a clinical study requiring administration of an investigational product (ie, not yet marketed), including expanded access or compassionate use

  * Exceptions:

    * Administration of investigational product with emergency use authorization granted for treatment of COVID 19 (eg, remdesivir) is permitted
    * Convalescent plasma as part of approved special access programs such as expanded access, emergency IND, or compassionate use is permitted
* Pregnant or breastfeeding (female subjects)
* Intubated and requires mechanical ventilation (including ECMO) at time of randomization

  * Exception: use of HFNC oxygen and noninvasive ventilation are permitted
* Endotracheal intubation is imminent, in the opinion of the investigator
* Not expected to survive for more than 48 hours after hospital admission, in the opinion of the investigator
* Presence of any of the following comorbid conditions before randomization and prior to SARS-CoV-2 infection:

  * New York Heart Association class IV heart failure
  * Stage 4 or 5 chronic kidney disease or requires renal replacement therapy
  * Biopsy proven cirrhosis, portal hypertension or hepatic encephalopathy
  * Stage IV malignancy
  * Chronic lung disease requiring home oxygen
  * Active tuberculosis
* History or evidence of pulmonary alveolar proteinosis
* Confirmed diagnosis or clinical suspicion of bacterial pneumonia or active uncontrolled bacterial, fungal, or non SARS-CoV-2 viral infection at Screening
* Absolute neutrophil count (ANC) value < 5 × 109 cells/L at Screening (can be lowered up to < 1.5 × 109 cells/L after Independent Data Monitoring Committee review of safety data, if CSL324 induced neutropenia is not assessed as a safety concern)
* Currently receiving a prohibited therapy including G-CSF, granulocyte-macrophage colony-stimulating factor (GM-CSF), or antibody against interleukin 6 (IL-6) / IL 6 receptor (anti IL-6 / 6R)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects progressing to endotracheal intubation or death prior to endotracheal intubation | Randomization to Day 28

SECONDARY OUTCOMES:
Proportion of deaths from all causes | Randomization to Day 28
Proportion of subjects intubated | Randomization to Day 28
Median length of stay in hospital | Randomization to Day 28
Number and proportion of subjects with at least a 2-point improvement in the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale | Randomization to Day 28
Number and proportion of subjects within each of the categories of the NIAID ordinal scale | Daily up to Day 28
Proportion of subjects using continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) | Randomization to Day 28
Proportion of subjects using high-flow nasal cannula (HFNC) | Randomization to Day 28
Proportion of subjects using extracorporeal membrane oxygenation (ECMO) | Randomization to Day 28
Maximum Change in Sequential Organ Failure Assessment (SOFA) score | Randomization to Day 28
Change in SOFA score and in individual components of the SOFA score | Baseline to Day 28
Number and proportion of subjects experiencing adverse events (AEs) | Up to 60 days
Number and proportion of subjects experiencing serious adverse events (SAEs) | Up to 60 days
Number and proportion of subjects experiencing adverse events of special interest (AESIs) | Up to 60 days
Presence of anti-CSL324 antibodies | Up to 28 days
Maximum concentration (Cmax) of CSL324 | Up to 28 days
Time to reach maximum concentration (Tmax) of CSL324 | Up to 28 days
Area under the concentration-time curve (AUC0-last) of CSL324 | Up to 28 days
Trough concentration (Ctrough) of CSL324 | Before dose on Day 4 and Day 8

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.